CLINICAL TRIAL: NCT03588780
Title: PREDICTEURS ET IMPACT CLINIQUE DE LA THROMBOSE DU STENT APRES LES THROMBECTOMIES CEREBRALES POUR LES OCCLUSIONS EN TANDEM
Brief Title: Stent Thrombosis After Tandem Lesions Thrombectomy
Acronym: DST-TANDEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7167
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-07

CONDITIONS: Acute Stroke With Large Vessel Occlusion
Keywords: acute stroke; thrombectomy; tandem lesions
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to describe the rate of delayed stent thrombosis after endovascular management of consecutive tandem lesions, in a patient series with systematic follow-up of stent patency. In addition, Investigatros aim to research baseline patient characteristics that are associated with a higher risk of delayed stent thrombosis and to evaluate the clinical consequences of stent thrombosis

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endovascular treatments for acute ischemic stroke in Strasbourg University Hospitals between 01/01/2009 and 01/04/2018
* Association of extracranial internal carotid artery (ICA) occlusion or stenosis ≥70% using NASCET criteria and an intracranial arterial occlusion in the anterior circulation

Exclusion Criteria:

- Endovascular treatments for complication of surgical carotid endarterectomy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent endovascular treatments for acute ischemic stroke in Strasbourg University Hospitals between 01/01/2009 and 01/04/2018
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Stent thrombosis rate | participants will be followed for the duration of hospital stay, an expected average 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Rémy BEAUJEUX, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Neuroradiologie Interventionnelle, Strasbourg, France